CLINICAL TRIAL: NCT05413291
Title: Natural History Protocol for Movement Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000865; 000865-N
Record Dates: First submitted 2022-06-09; First posted 2022-06-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11-07

CONDITIONS: Movement Disorder; Tremor; Parkinson's Disease
Keywords: Movement Disorder; Tremor; Parkinson's Disease; Natural History
MeSH Terms: conditions — Movement Disorders; Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- family members: family members who are 2 years old or older of people with movement disorders
- patients: subjects with movement disorders who are 2 years old or older

SUMMARY:
Background:

A movement disorder is a condition that causes a person s body to move in ways that are not normal. There are different types. Some disorders cause movements people can t control, such as tics or shaking. Some cause reduced or slow movements. Movement disorders can cause disability in people. Sometimes members of the same family will have the same disorder. Researchers want to learn more about how people develop these disorders. This research could lead to better treatments.

Objective:

This natural history study will collect data on people with different types of movement disorders. It will also collect data on their family members. The data will support further research.

Eligibility:

Children and adults aged 2 years and older who have a movement disorder. Family members of people with movement disorders are also needed.

Design:

Participants will undergo screening. They will have a physical exam. Researchers will look at their existing medical images. Any photographs or videos of their movements will also be reviewed.

Most participants will come to the NIH clinic for only 1 visit. They will answer questions about their condition. They will have normal tests used to diagnose their condition. They may have blood tests and different types of imaging scans. They may have tests to see how well their nerves function. The tests used will depend on the type of disorder they have.

Family members will have some of the same tests as people with disorders.

Participants will not receive any new treatments.

Some participants may be asked to return for a follow-up visit.

Up to 4000 people may participate.

DETAILED DESCRIPTION:
Study Description:

This is a Natural History and Screening protocol for movement disorders, no research procedures will be done but the resulting data will be used for research.

Objectives:

Primary Objective: To collect data as part of standard of care evaluation of patients who have or are suspected to have a movement disorder and their family members for use in future secondary research.

Endpoints:

Collection of data from clinical/routine care that will contribute to/be used for future research.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 2 and above
* Either one of these:

  * Have or suspected to have a diagnosis of a movement disorder.
  * Family member of someone who has or is suspected of having a diagnosis of a movement disorder.
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets the following criteria will be excluded from participation in this study:

-Being < 2 years old.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The following population groups may participate: - Subjects with neurological disorders who are 2 years old or older, - Family members who are 2 years old or older of people with a neurological disorder
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
to screen patients with movement disorders and family members of patients with movement disorders for enrollment in additional research protocols | throughout protocol
  The goal is to screen patients with movement disorders and family members of patients with movement disorders for enrollment in additional research protocols. No investigational treatments will be administered on this protocol and the NIH physicians will be playing a consultative role to the patient s primary physician.

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD stored in the database will be shared.
Supporting Information: Study Protocol
Time Frame: Data will be shared no later than 1 year after the last patient visit and data will be shared for at least 2 years.
Access Criteria: We do plan on broad data sharing. Therefore, there will be no restrictions on whom the de-identified data can be shared with.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000865-N.html